CLINICAL TRIAL: NCT04306029
Title: Improving Adherence to Postpartum Family Planning Guidance in Ghana: a Hybrid Type 2 Implementation and Effectiveness Study
Brief Title: Improving Adherence to Postpartum Family Planning Guidance in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: World Health Organization (Other); University of Ghana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 834804
Record Dates: First submitted 2020-03-05; First posted 2020-03-12 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Contraception

STUDY DESIGN:
Intervention Model Description: Hybrid Type II implementation and effectiveness study using a quasi-experimental stepped-wedge design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Intervention (No Intervention)
- Post-Intervention (Experimental): Postpartum staff has received the "Postpartum Family Planning Package," which consists of provider education on contraceptive delivery in the immediate postpartum period and promotion of the WHO MEC/PFP Compendium mobile application.
  Interventions: Other: Postpartum Family Planning Package

INTERVENTIONS:
Other: Postpartum Family Planning Package — "Postpartum Family Planning Package," which consists of provider education on contraceptive delivery in the immediate postpartum period and promotion of the WHO MEC/PFP Compendium mobile application.
  Arms: Post-Intervention

SUMMARY:
Evaluating a Postpartum Family Planning Package (PPFP) in a Hybrid Type II implementation study with a stepped-wedge design.

DETAILED DESCRIPTION:
Our overarching goal is to enable providers to consistently offer and deliver highly effective postpartum family planning methods in accordance with international guidelines. Our primary objective in this research is to assess the implementation and effectiveness of the "Postpartum Family Planning Package (PFPP)," an implementation strategy that consists of the following components: 1) a provider training on contraceptive methods available in the immediate postpartum period, and techniques for their placement in the case of intrauterine devices and implants, with quarterly booster trainings, and 2) promotion of the WHO MEC/Postpartum Family Planning Compendium mobile application as a provider decision tool to aid in postpartum family planning counselling.

ELIGIBILITY:
Provider Inclusion Criteria:

* Providers who care for postpartum women on the inpatient postpartum ward, including midwives, nurses, residents, fellows, and consultant physicians.

Provider Exclusion Criteria:

* Students caring for postpartum patients on the postpartum ward.

Client Inclusion Criteria:

- Women receiving antenatal care who have the potential to be admitted to the inpatient postpartum ward following delivery, or women admitted in the postpartum ward.

Client Exclusion Criteria:

- None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2142 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Provider discussed all guideline-appropriate contraceptive methods as defined by World Health Organization Medical Eligibility Criteria (yes/no) | During postpartum inpatient stay, prior to hospital discharge (approximately 2 days)

CONTACTS AND LOCATIONS:
Locations (3):
- Ghana (3):
  - Nsawam Goverment Hospital, Nsawam, Eastern Region
  - Ga West Municipal Hospital, Amasaman, Greater Accra Region
  - Maamobi Hospital, Accra

IPD SHARING:
Plan to Share IPD: No